CLINICAL TRIAL: NCT06593002
Title: The Effect of Pre-Treatment Therapeutic Play With Nursing Students on Children's Pain and Fear and on the Satisfaction Levels of Parents and Students
Brief Title: The Effect of Therapeutic Play on Children's Pain and Fear and Parents and Students' Satisfaction Levels
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Sibel Küçükoğlu, Prof, Selcuk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: SelcukUni2525
Record Dates: First submitted 2024-09-06; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Child Behavior; Pain; Anxiety; Anxiety and Fear
Keywords: Pain; Anxiety; Children; Nursing Student; therapeutic play
MeSH Terms: conditions — Child Behavior; Pain; Anxiety Disorders | interventions — Play Therapy

STUDY DESIGN:
Intervention Model Description: The universe of the study consisted of hospitalized children aged 3-6, their primary caregivers, and 3rd year nursing students taking the Pediatric Nursing course.
  Children and Parents: G*Power 3.1.9.6. program was used to calculate the sample size of the study. According to the a priori power analysis of the study with one-way hypothesis, 0.634 effect size, 0.05 significance level, and 0.80 power; it was determined that including a total of 64 (Experiment: 32 children + parents, Control: 32 children + parents) children in the study would provide a sufficient sample size.
  Nursing students: No sample calculation method was used, and all students who wanted to make therapeutic toys and play games with their patients were included in the study. 141 students who wanted to participate in the study out of a total of 178 students taking the course were included in the study.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Therapeutic play (Experimental): Children in the experimental group received a therapeutic video game intervention in addition to the pre-treatment routine.
  Interventions: Behavioral: Therapeutic play
- Control group (No Intervention): Children in the control group underwent routine clinical practice. No other intervention was performed.

INTERVENTIONS:
Behavioral: Therapeutic play — The children in the experimental group were given a therapeutic toy designed for them by the student nurse half an hour before the treatment, the toy and game were introduced, and they were allowed to play with this toy for half an hour, accompanied by the student nurse.
  Arms: Experimental: Therapeutic play

SUMMARY:
This study aims to determine the effects of playing with therapeutic toys made by nursing students on children's fear and pain levels towards treatment and the satisfaction levels of student nurses and parents.

DETAILED DESCRIPTION:
There are a limited number of studies in the literature examining the effects of therapeutic play implemented by nursing students. Although there are many studies showing that therapeutic play intervention is an effective intervention for sick children, it is seen that these studies are mostly conducted by researchers or clinical staff, and nursing students who have been in pediatric wards for a long time due to their clinical practices are far from therapeutic play practices. Therapeutic play may be a way for nursing students to initiate communication with children more easily. Therefore, there is a need for large-scale studies including nursing students. Starting from their student years, nursing students using therapeutic play as a means of communication with sick children may make them more willing to use such activities in their professional lives. In addition, determining the satisfaction levels is important for the continuation of such studies in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Having a child aged 3-6
* Having at least two days of inpatient treatment in the hospital (to gain experience with medication administration)
* Being accompanied by a parent
* Having one invasive drug treatment ordered by a doctor - Knowing and speaking Turkish
* Being willing to participate in the study

Exclusion Criteria:

* Those who are in intensive care,
* Those who have undergone surgery,
* Those who do not have a companion with their mother,
* Children with neurological and psychological disorders and parents,
* Children who only receive oral medication (as the level of pain and fear related to treatment will be low)

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 64 (Actual)
Dates: Start 2022-04-15 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2022-12-15 (Actual)

PRIMARY OUTCOMES:
Child and Parent Information Form | First measurement: 30 minute before treatment
  This form, developed by the researcher in line with the literature, was created to determine the descriptive characteristics of children and parents receiving inpatient treatment. This form was filled out by the parents of the children receiving inpatient treatment, using a face-to-face interview technique, half an hour before the treatment.
Wong-Baker Pain Scale | First measurement: Just before treatment
  It was developed by Wong and Baker in 1988. Patients' pain levels are evaluated by numbering their facial expressions. The numbering is as follows; "0" No pain, "1" A little pain, "2" A little more, "3" A lot more, "4" Quite a lot, "5" The most severe pain level. An increase in the score indicates that the severity of the pain also increases. This form was filled just before treatment.
Child Fear Scale | First measurement: Just before treatment
  It was developed by McMurtry and his colleagues to measure the fear levels of children aged 4-10. The scale is used to measure the child's fear level. The CQ is a scale that evaluates between 0-4, consisting of five drawn facial expressions ranging from a neutral expression (0=no fear) to a frightened face (4=severe fear). This form was filled just before treatment.

SECONDARY OUTCOMES:
Wong-Baker Pain Scale | Second measurement: within five minutes after the treatment is completedAfter treatment
  It was developed by Wong and Baker in 1988. Patients' pain levels are evaluated by numbering their facial expressions. The numbering is as follows; "0" No pain, "1" A little pain, "2" A little more, "3" A lot more, "4" Quite a lot, "5" The most severe pain level. An increase in the score indicates that the severity of the pain also increases. This form was measured a second time immediately after treatment.
Child Fear Scale | Second measurement: within five minutes after the treatment is completed
  It was developed by McMurtry and his colleagues to measure the fear levels of children aged 4-10. The scale is used to measure the child's fear level. The CQ is a scale that evaluates between 0-4, consisting of five drawn facial expressions ranging from a neutral expression (0=no fear) to a frightened face (4=severe fear). This form was measured a second time immediately after treatment.
Student Satisfaction Survey | Within five minutes after the treatment is completed
  The form prepared by the researchers specifically asked about the student nurses' satisfaction with making toys and playing with the sick child. It was filled out by the student nurses after the treatment.
Parent Satisfaction Survey | Within five minutes after the treatment is completed
  The form prepared by the researchers specifically asked about parents' satisfaction with student nurses making toys and playing games for their children. It was filled out by parents after the treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Sibel Küçükoğlu, Study Director — Selcuk University
Locations (1):
- Selcuk University, Konya, Selcuklu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
It can be shared after publication.

REFERENCES:
- [Result] Inan G, Inal S. The Impact of 3 Different Distraction Techniques on the Pain and Anxiety Levels of Children During Venipuncture: A Clinical Trial. Clin J Pain. 2019 Feb;35(2):140-147. doi: 10.1097/AJP.0000000000000666. PMID 30362982
- [Result] Gates M, Hartling L, Shulhan-Kilroy J, MacGregor T, Guitard S, Wingert A, Featherstone R, Vandermeer B, Poonai N, Kircher J, Perry S, Graham TAD, Scott SD, Ali S. Digital Technology Distraction for Acute Pain in Children: A Meta-analysis. Pediatrics. 2020 Feb;145(2):e20191139. doi: 10.1542/peds.2019-1139. Epub 2020 Jan 22. PMID 31969473
- [Result] Li WHC, Chung JOK, Ho KY, Kwok BMC. Play interventions to reduce anxiety and negative emotions in hospitalized children. BMC Pediatr. 2016 Mar 11;16:36. doi: 10.1186/s12887-016-0570-5. PMID 26969158